CLINICAL TRIAL: NCT00124423
Title: Megavoltage CT (MVCT) Imaging for Intracavitary Radiation Treatment in Cervix Cancer
Status: Completed | Type: Observational
Sponsor: AHS Cancer Control Alberta (Other)
Responsible Party: Sponsor
Other Study IDs: GY-03-0018/ethics 21373
Record Dates: First submitted 2005-07-26; First posted 2005-07-28 (Estimated); Last update posted 2016-02-26 (Estimated); Status verified 2012-04

CONDITIONS: Cervix Cancer
Keywords: brachytherapy megavoltage CT imaging
MeSH Terms: conditions — Uterine Cervical Neoplasms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Procedure: Megavoltage CT scan

SUMMARY:
The Cross Cancer Institute has recently acquired a tomotherapy radiotherapy treatment machine; the first of its kind in Canada. It has the potential to improve cancer treatment outcomes where radiotherapy is used. Cervix cancer is a disease where radiotherapy is a particularly important treatment modality. The researchers believe that by combining tomotherapy (which has the ability to give higher doses of radiation to areas of cancer while sparing normal tissues) with radiotherapy given from inside the uterus and vagina (brachytherapy) disease outcomes will be improved. For this to be possible the researchers will need to accurately map the doses of radiation given to the cervix, uterus and other pelvic organs from these two types of radiation treatment. As well as being used for treatment, the tomotherapy machine can also be used for taking medical images by using very much lower doses of radiation. This study will allow the researchers to develop the mapping process by using very low doses of radiation on the tomotherapy unit to take medical x-ray images of patients being treated by brachytherapy for cervix cancer. In this special circumstance the researchers expect the images to be of a higher quality than for conventional computed tomography (CT) scanning or magnetic resonance imaging (MRI) scanning.

DETAILED DESCRIPTION:
Megavoltage CT Imaging for Intracavitary Radiation Treatment in Cervix Cancer

Proposal

To assess the feasibility of performing CT imaging using a megavoltage CT scanner on five patients where remote afterloading intracavitary applicators have been inserted for the purpose of delivering intracavitary radiotherapy in the treatment of cervix cancer.

Rationale

While there has been recent improvements in the treatment of more advanced stages of cervix cancer by combining radical radiation treatment with concurrent cisplatin based chemotherapy, there is room for further improvements in local regional control. One approach to achieving this is to increase the dose of therapeutic radiation to the clinical target volume without exceeding the tolerance of the adjacent normal tissues. Modern radiotherapy techniques allow for better conformation of the high dose radiation volume to the clinical target volume by using external beam techniques (conformal radiation treatment and intensity modulated radiation treatment) and the use of tomotherapy is likely to be particularly advantageous in this regard. The mainstay of cervix cancer radiotherapy has always been and will likely remain the use of brachytherapy. Future improvements in the outcome of cervix cancer treated by radiotherapy are therefore likely to necessitate accurately combining intracavitary radiation treatment with intensity modulated external beam radiation treatment and particularly with the use of tomotherapy techniques.

The ability to accurately reconstruct the three-dimensional dosimetry achieved by the combined use of intracavitary radiation treatment and helical tomotherapy will be pivotal in the success of this strategy. Conventional CT imaging of patients receiving intracavitary radiation treatment is hampered by distortion artifacts from the metallic applicators. The opportunity to gain improved images using megavoltage CT scanning using the same equipment and same patient set-up that will ultimately by used for the delivery of tomotherapy offers some unique potential advantages and solutions to the problem.

By imaging patients with the remote afterloading applications in situ, the researchers should be able to generate accurate isodose distributions in three dimensions for the intracavitary component of the cervix cancer treatment. By contouring the clinical target volume, which includes the primary cancer, local routes of spread and regional pelvic lymph nodes, the researchers can explore the feasibility of generating combined helical tomotherapy and intracavitary radiation treatment plans.

Patients and Methods

Patients who are to receive intracavitary brachytherapy on the low dose rate selectron at the Cross Cancer Institute will be approached to participate in this pilot study. An informed consent will be obtained from five patients for this study. Following the insertion of the remote afterloading applicators in the operating room, patients are normally transferred from the operating room to Simulator C for orthogonal simulator films and then to Station 30 where treatment is started approximately two hours later after dosimetry calculations have been performed and treatment has been prescribed.

For the patients consenting to this study, they will proceed from Simulator C to Station 30 via the tomotherapy unit in CBIAR where megavoltage CT scans will be taken. Patients will be accompanied by a brachytherapy radiation therapist. The megavoltage CT scans will take approximately one hour to perform, but this will not result in any treatment delay for the patient.

Isodose volumes from the prescribed intracavitary brachytherapy will be reconstructed on the megavoltage images. The feasibility of defining the clinical target volume on the megavoltage scans will be explored. This may require fusion with conventional CT images that will already have been taken for diagnostic and external beam treatment planning purposes. Megavoltage and/or fused images will be used to pilot the integration of tomotherapy intensity modulated radiation therapy treatment plans with intracavitary brachytherapy dosimetry.

The current study will have no influence on individual patient treatments but is a prelude to a potential dose escalation study using tomotherapy for patients with cervix cancer.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing brachytherapy for cervix cancer

Exclusion Criteria:

* Patient refusal

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: community sample
Sampling Method: Non-Probability Sample
Enrollment: 5 (Actual)
Dates: Start 2004-06; Primary Completion 2007-06 (Actual); Study Completion 2007-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Robert Pearcey, MD, Principal Investigator — AHS Cancer Control Alberta
Locations (1):
- Cross Cancer Institute, Edmonton, Alberta, Canada